CLINICAL TRIAL: NCT04536948
Title: Which Cold Application is More Effective in Patients With Lateral Epicondylitis?
Brief Title: Cold Application in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nihan Ozunlu Pekyavas, Associated Proffesor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA16 / 369
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Lateral Epicondylitis
Keywords: Kinesio Tape; Thermal Analysis; Cold
MeSH Terms: conditions — Tennis Elbow; Common Cold | interventions — methyl salicylate

STUDY DESIGN:
Intervention Model Description: Fifty-four volunteers diagnosed with lateral epicondylitis were included in our study and were randomly divided into two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Cooling gel application
  Interventions: Other: Cooling Gel
- Group 2 (Active Comparator): Cold pack was applied
  Interventions: Other: Cold Pack

INTERVENTIONS:
Other: Cooling Gel — Cooling gel (Nelsons Arnicare Arnica Cooling Gel) was applied to the lateral epicondyle region with sponge head 3 times a day. The cooling gel was applied to the painful area around the lateral epicondyle
  Arms: Group 1
Other: Cold Pack — Cold pack was applied to the painful area for 15 minutes on a moist towel placed on the painful area around the lateral epicondyle.
  Arms: Group 2

SUMMARY:
Purpose: The purpose of this study was to investigate which cold application is more effective to regulate skin temperature in patients with lateral epicondylitis. Materials and Methods: Fifty-four patients with lateral epicondylitis were randomly divided into 2 groups as cooling gel (n=27) group and cold pack (n=27) group. Cooling gel and cold pack applications were applied on painful lateral epicondyle region for 15 minutes. Patients were assessed before and after the application. Assessments included the severity of pain during wrist extension, evaluated by Visual Analog Scale (VAS) and thermal imaging of lateral epicondyle region evaluated by Infrared Thermography (FLIR5 Thermal Camera).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with elbow pain for at least 3 months
* those between 20 and 40 years of age
* who did not have cold allergies

Exclusion Criteria:

* With a different elbow problem or multiple elbow problems,
* having cervical or other upper extremity problems,
* elbow joint operation,
* tendon rupture,
* limited range of motion due to humerus, radius or ulna fracture
* individuals with a history of osteoporosis, malignancy, hemophilia, neurological effect, and cognitive dysfunction

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Pain Severity | 15 minutes
  The severity of shoulder pain at rest, night and activity was evaluated by Visual Analogue Scale (VAS). Accordingly, in a line of 10 cm 0 point refers to no pain, 10 point was considered to be the maximum value of pain. Patients were asked to mark the severity of their pain and tape measurement was recorded in cm.
Thermographic Assessment | 15 minutes
  Infrared thermography (IRT) uses a thermal camera that receives and processes the infrared radiation emitted from the surface of the body. Thus, IRT records the temperature distribution of the skin.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No